CLINICAL TRIAL: NCT02521428
Title: End-of-Life Decisions in Surgical Intensive Care Medicine - The Relevance of Treatment Withholding
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jan Adriaan Graw, Dr. med., Charite University, Berlin, Germany
Other Study IDs: EOLD_T
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: retrospective analysis — Approximately 200 patients will be enrolled in the study. They are followed up until their death on the ICU. In clinical routine end-of-life decisions are documented for decision-makers and procedures in the patients´ records. Patients´ characteristics and therapeutic approaches are documented in the electronic patient data management system.

SUMMARY:
The purpose of this retrospective observational study is to describe the sequence of ICU-therapies that are limited and to compare characteristics and the decision making process in surgical ICU-patients.

DETAILED DESCRIPTION:
Decisions to limit life-support therapy are common on the intensive care unit (ICU). End-of-life decisions (EOLD) underlie a dynamic process and limitation of ICU-therapies is done sequentially. Questionnaire-based and observational studies on medical ICUs and in palliative care reveal blood transfusions as the first therapy physicians withhold in EOLDs. Whether this practice also applies to surgical ICU-patients is unknown.

The purpose of this retrospective observational study is to describe the sequence of ICU-therapies that are limited and to compare characteristics and the decision making process in surgical ICU-patients.

ELIGIBILITY:
Inclusion Criteria:

* All surgical patients admitted to the ICU All surgical patients discharged death from the ICU

Exclusion Criteria:

* All patients discharged alive from the ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Surgical Intensive Care Department patients will be enrolled in the study
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2008-08; Primary Completion 2011-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
sequence of withdrawing life-sustaining treatment | 3 years
  The primary objective of this study performed according to an observational post-ad-hoc design is to identify the sequence of withdrawing life-sustaining treatment in surgical ICU-patients with an end-of-life decision on an intensive care unit of a German academic medical center.
  Approximately 200 patients will be enrolled in the study. They are followed up until their death on the ICU. In clinical routine end-of-life decisions are documented for decision-makers and procedures in the patients´ records. Patients´ characteristics and therapeutic approaches are documented in the electronic patient data management system.

SECONDARY OUTCOMES:
factors associated with the withholding of specific ICU-therapies | 3 years
  Approximately 200 patients will be enrolled in the study. They are followed up until their death on the ICU. In routine end-of-life decisions are documented for decision-makers and procedures in the patients´ records. Patients´ characteristics and therapeutic approaches are documented in the electronic patient data management system